CLINICAL TRIAL: NCT03035279
Title: An Open Label Phase 1 Study of SC-006 as a Single Agent and in Combination With ABBV-181 in Subjects With Advanced Colorectal Cancer
Brief Title: A Study of SC-006 and in Combination With ABBV-181 in Subjects With Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M16-312
Record Dates: First submitted 2017-01-23; First posted 2017-01-30 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
Keywords: Advanced colorectal cancer; Cancer; Metastatic colorectal cancer; Unresectable colorectal cancer; Maximum tolerated dose; Pharmacokinetics
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (Experimental): SC-006 Dose regimen finding
  Interventions: Drug: SC-006
- Arm B (Experimental): SC-006 Dose expansion
  Interventions: Drug: SC-006
- Arm C (Experimental): SC-006 and ABBV-181 Combination escalation and expansion
  Interventions: Drug: SC-006; Drug: ABBV-181

INTERVENTIONS:
Drug: SC-006 — Intravenous
Drug: ABBV-181 — Intravenous
  Arms: Arm C

SUMMARY:
This is a multicenter, open-label, Phase 1 study of SC-006 given as a single agent and in combination with ABBV-181 in participants with advanced colorectal cancer (CRC), and consists of Part A (single agent SC-006 dose regimen finding), followed by Part B (single agent SC-006 dose expansion), and Part C (SC-006 and ABBV-181 combination escalation and expansion). Part A (dose regimen finding) will involve dose escalation and possible dose interval modification to define the maximum tolerated dose (MTD) and/or recommended Part B dose and schedule. Part B (dose expansion) will enroll additional participants who will be treated with a study drug dose at or below the MTD determined in Part A. Part C is dose escalation of SC-006 and fixed dose of ABBV-181 in combination. Recommended dose cohort of SC-006 with ABBV-181 will be expanded.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically confirmed advanced metastatic or unresectable colorectal cancer (CRC) that is relapsed, refractory, or progressive following at least 2 prior systemic regimens in the metastatic setting.
* Participants with an Eastern Cooperative Oncology Group (ECOG) of 0 - 1.
* Participants with adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

* Participants with prior exposure to a pyrrolobenzodiazepine or indolinobenzodiazepine based drug.

Additional Exclusion Criteria for the SC-006 and ABBV-181 Combination Treatment Regimen:

* History of inflammatory bowel disease
* Active autoimmune disease, with exception of psoriasis not requiring systemic treatment, vitiligo, type 1 diabetes mellitus and hypothyroidism
* History of primary immunodeficiency, allogenic bone marrow transplantation, solid organ transplantation, or previous clinical diagnosis of tuberculosis
* History of immune-mediated pneumonitis
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLT) | Minimum first cycle of dosing (21-day cycles)
  DLTs graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 2 years
  OS is defined as the time from the participant's first dose date to death due to any cause.
Progression Free Survival (PFS) | Approximately 2 years
  PFS time is defined as the time from the participant's first dose of study drug (Day 1) to either the participant's disease progression or death due to any cause.
Time to Cmax (Tmax) of SC-006 | Approximately 1 year
  Time to Cmax of SC-006
Area under the plasma concentration-time curve within a dosing interval (AUC) of SC-006 | Approximately 1 year
  Area under the plasma concentration-time curve within a dosing interval of SC-006
Duration of Clinical Benefit (DOCB) | Approximately 2 years
  DOCB is defined as the time from the initial partial response (PR), complete response (CR), or stable disease to disease progression.
Objective Response Rate (ORR) | Approximately 2 years
  ORR is defined as the percentage of participants whose best overall response is either complete response (CR) or partial response (PR), as determined by Investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Terminal half life (T1/2) of SC-006 | Approximately 1 year
  Terminal half life (T1/2) of SC-006
Duration of response (DOR) | Approximately 2 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to disease progression or death, whichever occurs first.
Observed plasma concentrations at trough (Ctrough) of SC-006 | Approximately 1 year
  Observed plasma concentrations at trough of SC-006
Clinical Benefit Rate (CBR) defined as CR, PR, or stable disease (SD) | Approximately 2 years
  CBR is defined as the percentage of participants who achieve a best response of CR, PR, or stable disease (SD).
Maximum observed serum concentration (Cmax) of SC-006 | Approximately 1 year
  Maximum observed serum concentration of SC-006

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (9):
- United States (9):
  - Highlands Oncology Group /ID# 201182, Fayetteville, Arkansas
  - University of California, Los Angeles /ID# 160882, Los Angeles, California
  - University of Michigan Hospitals /ID# 167101, Ann Arbor, Michigan
  - Mayo Clinic - Rochester /ID# 160884, Rochester, Minnesota
  - Washington University-School of Medicine /ID# 160883, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center /ID# 160881, New York, New York
  - Carolina BioOncology Institute /ID# 202712, Huntersville, North Carolina
  - Oklahoma University /ID# 202713, Oklahoma City, Oklahoma
  - Tennessee Oncology-Nashville Centennial /ID# 160880, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No